CLINICAL TRIAL: NCT01362517
Title: Assessment of the Immunogenicity and Safety of Quinvaxem Vaccine (DTwP-HepB-Hib) Against Diphtheria, Pertussis, Tetanus, Hepatitis B and Diseases Caused by H. Influenzae Among Healthy Vietnamese Children
Brief Title: Study of Quinvaxem for Vaccination Against Diphtheria, Pertussis, Tetanus, Hepatitis B and Diseases Caused by Haemophilus Influenzae Type B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QVX-V-C001
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Diphtheria; Pertussis; Tetanus; Hepatitis B; Haemophilus Influenzae Infections
Keywords: Vaccination; Immunisation; Virus; Diphtheria; Pertussis; Tetanus; Hepatitis B; Haemophilus Influenzae; Immunity
MeSH Terms: conditions — Diphtheria; Whooping Cough; Tetanus; Hepatitis B; Haemophilus Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quinvaxem (Experimental)
  Interventions: Biological: Quinvaxem

INTERVENTIONS:
Biological: Quinvaxem — A single dose (0.5 mL) of Quinvaxem contains:
  diphtheria antitoxin (>= 30 IU), tetanus antitoxin (>= 60 IU), whole-cell inactive pertussis bacteria (>= 4 IU), 10 mcg Hib oligosaccharide conjugate (approx. 25 mcg CRM197), 10 mcg Hepatitis B surface antigen
  One dose of Quinvaxem given at 2, 3 and 4 months of age

SUMMARY:
The aim of this study was to evaluate the immunogenicity and safety of the Quinvaxem vaccine (a liquid combination vaccine against diphtheria, tetanus, B. pertussis, hepatitis B and H. influenzae Type B). Healthy Vietnamese infants received three doses of vaccine at 2, 3 and 4 months of age according to the local Expanded Programme on Immunisation (EPI) schedule

ELIGIBILITY:
Inclusion Criteria:

* Infants are at age of DTP vaccination of the local EPI program (60-120 days old) and free from any obvious health problems
* Have a normal gestational age (≥ 37 weeks); birth weight > 2.5 kg
* There is no congenital disease detected through interview and clinical examination
* Already had or not yet received Hepatitis B vaccination at birth
* Do not have dermatological diseases such as eczema, allergies
* Parent or legal guardian voluntarily provides consent for their child for participation in the study by signing the informed consent and agrees to comply with all study procedures

Exclusion Criteria:

* Already vaccinated with DTP vaccine
* Have an acute infection at the time of study vaccination
* Contraindications to Quinvaxem
* Receiving treatment with systemic corticosteroids
* Currently participating in another clinical trial
* In receipt of a parenteral immunoglobulin preparation and/or blood/blood products since birth
* Parents intend to move to another location during the study (the next 12 months)

Ages: 60 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tran Ngoc Huu, PhD, MD, Principal Investigator — Pasteur Institute of Ho Chi Minh City
Locations (1):
- Pasteur Institute, Ho Chi Minh City, Vietnam

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in Vietnam First subject first visit (FSFV): April 2010 Last subject last visit (LSLV): April 2011
Groups:
- Quinvaxem: Quinvaxem : A single dose (0.5 mL) of Quinvaxem contains:
  diphtheria antitoxin (>= 30 IU), tetanus antitoxin (>= 60 IU), whole-cell inactive pertussis bacteria (>= 4 IU), 10 mcg Hib oligosaccharide conjugate (approx. 25 mcg CRM197), 10 mcg Hepatitis B surface antigen
  One dose of Quinvaxem given at 2, 3 and 4 months of age
Period: Overall Study
Arm/Group | Quinvaxem
Started | 131
Completed | 129
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Quinvaxem
Number analyzed (Participants) | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 131
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity - Seroprotection (Seroconversion for Pertussis) to Each Vaccine Component
Description: Assessment of the proportion of subjects who have seroconverted to each of the 5 vaccine components (D, T, P, HepB, Hib)
Time Frame: at 5 months (equivalent to 1 month after the third vaccination)
Population: Analysis population excludes one subject excluded as a protocol violator
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Quinvaxem
Number analyzed (Participants) | 130
percentage of subjects
  % of subjects with anti-diphtheria >=0.1 IU/mL | 93.1 [87.3 to 96.8]
  % of subjects with anti-pertussis >=20 EU/mL | 99.2 [95.8 to 100]
  % of subjects with anti-tetanus >=0.1 IU/mL | 98.5 [94.6 to 99.8]
  % of subjects with anti-hepatitis B >=10 mIU/mL | 93.1 [87.3 to 96.8]
  % of subjects with anti-PRP>=0.15 mcg/mL | 100 [97.2 to 100]

2. Primary Outcome: Immunogenicity - Seroprotection (Seroconversion for Pertussis) to Each Vaccine Component
Description: as for outcome 1
Time Frame: at 14 months (equivalent to 12 months after the first vaccination
Population: Analysis population excludes one subject excluded as a protocol violator and additionally at 14 months one lost to follow up
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Quinvaxem
Number analyzed (Participants) | 129
percentage of subjects
  % of subjects with anti-diphtheria >=0.1 IU/mL | 88.4 [81.5 to 93.3]
  % of subjects with anti-pertussis >=20 EU/mL | 49.6 [40.7 to 58.5]
  % of subjects with anti-tetanus >=0.1 IU/mL | 82.2 [74.5 to 88.3]
  % of subjects with anti-hepatitis B >=10 mIU/mL | 76.7 [68.5 to 83.7]
  % of subjects with anti-PRP >=0.15 mcg/mL | 97.7 [93.4 to 99.5]

3. Secondary Outcome: Safety: Adverse and Serious Adverse Events
Description: Assessment of the proportion of children with adverse events and/or serious adverse events following each Quinvaxem vaccine injection
Time Frame: From Day 1 up to 30 days after the third vaccination
Measure: Number; unit: Number of children with AE per 100 doses
Units Other Than Participants: Doses
Arm/Group | Quinvaxem
Number analyzed (Participants) | 131
Number analyzed (Doses) | 392
Number of children with AE per 100 doses
  Injection site swelling | 5.6
  Injection site redness | 2.8
  Injection site pain | 4.1
  Fever (>=38 deg C) | 18.4
  Rash | 0.3
  Loss of appetite | 2.6
  Vomiting | 1.0
  Diarrhea | 3.0
  Irritability | 7.9
  Abnormal crying | 0
  Persistent crying | 0.5
  Drowsiness | 0.5

ADVERSE EVENTS:
Time Frame: Parents of subjects recorded solicited local and systemic and unsolicited adverse events from baseline up to 28 days after vaccination.
Groups:
- First Dose: Quinvaxem : A single dose (0.5 mL) of Quinvaxem contains:
  diphtheria antitoxin (>= 30 IU), tetanus antitoxin (>= 60 IU), whole-cell inactive pertussis bacteria (>= 4 IU), 10 mcg Hib oligosaccharide conjugate (approx. 25 mcg CRM197), 10 mcg Hepatitis B surface antigen
  One dose given at 2 months of age
- Second Dose: Quinvaxem : A single dose (0.5 mL) of Quinvaxem contains:
  diphtheria antitoxin (>= 30 IU), tetanus antitoxin (>= 60 IU), whole-cell inactive pertussis bacteria (>= 4 IU), 10 mcg Hib oligosaccharide conjugate (approx. 25 mcg CRM197), 10 mcg Hepatitis B surface antigen
  One dose given at 3 months of age
- Third Dose: Quinvaxem : A single dose (0.5 mL) of Quinvaxem contains:
  diphtheria antitoxin (>= 30 IU), tetanus antitoxin (>= 60 IU), whole-cell inactive pertussis bacteria (>= 4 IU), 10 mcg Hib oligosaccharide conjugate (approx. 25 mcg CRM197), 10 mcg Hepatitis B surface antigen
  One dose given at 4 months of age
Arm/Group | First Dose | Second Dose | Third Dose
Serious Adverse Events (participants affected / at risk) | 4/131 | 6/131 | 1/130
Other Adverse Events (participants affected / at risk) | 75/131 | 34/131 | 25/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Dose (N=131) | Second Dose (N=131) | Third Dose (N=130)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Dose (N=131) | Second Dose (N=131) | Third Dose (N=130)
Pyrexia (General disorders) | 34 (34) | 20 (20) | 18 (18)
Feeding disorder (Metabolism and nutrition disorders) | 10 (10) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 5 (5)
Irritability (Psychiatric disorders) | 21 (21) | 8 (8) | 2 (2)
Injection site induration (General disorders) | 19 (19) | 3 (3) | 0 (0)
Injection site erythema (General disorders) | 7 (7) | 2 (2) | 2 (2)
Injection site pain (General disorders) | 24 (24) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Persistent crying (General disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator to submit all manuscripts/abstracts to the sponsor for review at least 60 days prior to any intended submission.